CLINICAL TRIAL: NCT04020653
Title: A Pilot, Double-blind, Randomized, Parallel-group, Placebo-controlled, Exploratory Study to Assess the Safety and Efficacy of 5-aminolevulinic Acid Hydrochloride (5-ALA HCl) and Sodium Ferrous Citrate (SFC) Added on Artemisinin-based Combination Therapy (ACT) in Adult Patients With Uncomplicated Malaria
Brief Title: A Study to Assess the Safety and Efficacy of 5-aminolevulinic Acid Hydrochloride (5-ALA HCl) and Sodium Ferrous Citrate (SFC) Added on Artemisinin-based Combination Therapy (ACT) in Adult Patients With Uncomplicated Malaria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Considering the Thai FDA requirement, changes of Malaria cases in Thailand and EC recommendation, the decision to withdrawal the study was made.
Sponsor: Neopharma Japan Co., Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPJ005-MAL-0122
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Malaria
Keywords: Uncomplicated malaria; sodium ferrous citrate (SFC); 5-aminolevulinic acid hydrochloride (5-ALA HCl); artemisinin-based combination therapy
MeSH Terms: conditions — Malaria | interventions — Aminolevulinic Acid; ferrous citrate; Sodium Glutamate; Artemether; Lumefantrine; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo + ACT (Placebo Comparator): Patients will receive placebo for Day 1 to Day 7 and ACT (as per package instruction) for Day 1 to Day 3.
  Interventions: Drug: Artemisinin-based combination (ACT); Drug: Placebo
- 5 ALA/SFC+placebo+ACT BID (Experimental): 5-ALA HCl 300 mg and SFC 236 mg will be administered BID for Day 1 to Day 7 and ACT (as per package instruction) for Day 1 to Day 3.
  Patients will receive 5-ALA HCl+Placebo and SFC+Placebo at odd number of study medication dosing (Dose 1, 3, 5, 7, 9, 11, 13) and only 5-ALA HCl and SFC at even numbers of study medication dosing (Dose 2, 4, 6, 8, 10,12, 14).
  Interventions: Drug: Artemisinin-based combination (ACT); Drug: Placebo; Drug: 5-aminolevulinic acid hydrochloride (5-ALA HCl) 300 mg BID; Drug: Sodium ferrous citrate (SFC) 236 mg BID
- 5-ALA/SFC+placebo+ACT QD (Experimental): 5-ALA HCl 600 mg and SFC 472 mg will be administered QD in the morning or evening for Day 1 to Day 7 and ACT (as per package instruction) for Day 1 to Day 3. Patients will receive 5-ALA HCl and SFC at odd number of study medication dosing (Dose 1, 3, 5, 7) and placebo at even numbers of study medication dosing (Dose 2, 4, 6).
  Interventions: Drug: 5-aminolevulinic acid hydrochloride (5-ALA HCl) 600 mg QD; Drug: Sodium ferrous citrate (SFC) 472 mg QD; Drug: Artemisinin-based combination (ACT); Drug: Placebo

INTERVENTIONS:
Drug: 5-aminolevulinic acid hydrochloride (5-ALA HCl) 600 mg QD — 5-ALA HCl 150 mg capsules will be given to the patients as 600 mg QD
  Arms: 5-ALA/SFC+placebo+ACT QD
Drug: Sodium ferrous citrate (SFC) 472 mg QD — SFC 118 mg capsules will be given to the patients as 472 mg QD
  Arms: 5-ALA/SFC+placebo+ACT QD
Drug: Artemisinin-based combination (ACT) — Tablets of ACT will be administered following Dosage and Administration in the package insert of ACT. ACT will be supplied as a combination tablet.
  Other Names: Artemether 20 mg and lumefantrine 120 mg
Drug: Placebo — Matching placebo capsules to 5-ALA HCl and SFC will be administered to the patients
Drug: 5-aminolevulinic acid hydrochloride (5-ALA HCl) 300 mg BID — 5-ALA HCl 150 mg capsules will be given to the patients as 300 mg BID
  Arms: 5 ALA/SFC+placebo+ACT BID
Drug: Sodium ferrous citrate (SFC) 236 mg BID — SFC 118 mg capsules will be given to the patients as 236 mg BID
  Arms: 5 ALA/SFC+placebo+ACT BID

SUMMARY:
This is a pilot, double-blind, randomized, parallel-group, placebo-control, exploratory study to evaluate the efficacy and safety of 5-aminolevulinic acid hydrochloride (5-ALA HCl) and sodium ferrous citrate (SFC) added on artemisinin-based combination therapy (ACT) compared with ACT alone in the treatment of malaria. Patients who are suffering from uncomplicated malaria, are eligible for randomization.The study will be conducted in a total of 75 patients with uncomplicated malaria.

DETAILED DESCRIPTION:
Approximately 75 patients will be randomized in a 1:2:2 ratio to 3 arms:

Arm 1: placebo+ACT group (15 patients)

Arm 2: 5 ALA/SFC+Placebo+ACT twice daily (BID) (30 patients)

Arm 3: 5-ALA/SFC+Placebo+ACT once daily (QD) (30 patients)

The study duration will be a maximum of 98 days with treatment period of 7 days and follow-up period of 91 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of 18 to 60 years inclusive.
2. Weighing 35 to 90 kg.
3. Women with child bearing potential willing to give consent for pregnancy test.
4. Presence of symptomatic uncomplicated malaria of all species inclusive with a diagnosis confirmed by:

   A. Microscopically confirmed parasite infection, between 500 and 100,000 asexual parasite count/μL of blood.

   B. Fever, as defined by axillary/tympanic of ≥37.5°C within 24 hours before randomization (must be documented).
5. Patients must be willing and able to give written informed consent and comply with all study visits and procedures. If a patient cannot read informed consent and/or write a signature, an impartial witness who speaks the language of the patient must be present during the entire informed consent process and discussion with the patient.

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment according to the World Health Organization (WHO) Criteria 2010.
2. Severe vomiting, defined as more than three times in the 24 hours prior to inclusion in the study or inability to tolerate oral treatment.
3. Known history of photo-hypersensitivity, porphyria, or hemochromatosis.
4. Have taken any medication with antimalarial or antibiotic with antimalarial effect within 14 days before randomization.
5. Received an investigational drug within the past 28 days.
6. Patients whose Hemoglobin (Hb) level is lower than 8 g/dL.
7. Liver function tests (aspartate aminotransferase/alanine aminotransferase [AST/ALT] levels) more than 2.5 times upper limit of normal values.
8. Known human immunodeficiency virus (HIV) or Hepatitis C virus (HCV) or hepatitis B surface antigen (HBsAg) positive, testing is not required.
9. Known significant renal impairment as indicated by serum creatinine of ≥1.4 mg/dL or estimated glomerular filtration rate (eGFR) of <45 mL/min.
10. Known history of hypersensitivity, allergic or adverse reactions to 5-aminolevulinic acid and sodium ferrous citrate.
11. Presence or history of uncontrolled systemic disease.
12. Female patients who are pregnant or breast-feeding.
13. Any other condition in the opinion of the investigator makes the patient unsuitable for study
14. Received any medication specified as contraindication for ACT or affecting blood concentration of ACT within 5 times the half-life of each medication before the first dose of study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-06 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | From screening visit (Day -1) untill the Follow-up Visit (Day 98)
  Number of patients with any adverse events or clinically significant abnormal laboratory parameters to investigate safety and tolerability of 5-ALA HCl and SFC in simultaneous administration with ACT.
Cure rate on Day 28 | Day 28
  Cure rate is defined as the proportion of patients with polymerase chain reaction (PCR)-corrected Adequate Clinical and Parasitological Response (ACPR). PCR-corrected ACPR is defined as patients with clearance of asexual parasites within 28 days of initiation of study medication and without recrudescence within 28 days. Cure rate to investigate the preliminary efficacy of 5-ALA HCl and SFC in simultaneous administration with ACT.
Parasite Clearance Time | Every 4 hours for 72 hours from Day 1 to Day 7 until 4 consecutive negative readings
  Time from first dosing to time of first of 4 consecutive readings with zero parasite count in blood. Calculated based on parasite count in blood every 4 hours after the start of study medication for 72 hours until there are 4 consecutive negative readings.
Fever Reduction Time | Every 4 hours for 72 hours from Day 1 to Day 7
  Time to Fever Reduction is defined as the time from first dosing to first normal reading of temperature (<37.5 °C) for two consecutive normal temperature reading plus confirmed normal temperature every 4 hours after the start of study medication for 72 hours
Gametocyte Clearance Time | Day 1 to Day 7 + 24 hours
  Time from the first dose until first total and continued disappearance of gametocytes which remains at least a further 24 hours
Change in inflammatory parameter: C-reactive protein | Days 1, 3, 7, and 28
  Change from baseline in C-reactive protein to investigate change in inflammatory parameters
Change in inflammatory parameter: interleukin-6 | Days 1, 3, 7, and 28
  Change from baseline in interleukin-6 to investigate change in inflammatory parameters
Change in inflammatory parameter: tumor necrosis factor (TNF)-alpha | Days 1, 3, 7, and 28
  Change from baseline in tumor necrosis factor (TNF)-alpha to investigate change in inflammatory parameters
Change in iron metabolism: Serum iron | Days 1, 3, 7, 28, and 98
  Change from baseline in serum iron to investigate change in iron metabolism parameters
Change in iron metabolism: Hepcidin | Days 1, 3, 7, 28, and 98
  Change from baseline in hepcidin to investigate change in iron metabolism parameters
Change in iron metabolism: total iron binding capacity (TIBC) | Days 1, 3, 7, 28, and 98
  Change from baseline in total iron binding capacity (TIBC) to investigate change in iron metabolism parameters
Change in iron metabolism: unsaturated iron binding capacity (UIBC) | Days 1, 3, 7, 28, and 98
  Change from baseline in unsaturated iron binding capacity (UIBC) to investigate change in iron metabolism parameters

IPD SHARING:
Plan to Share IPD: Undecided